CLINICAL TRIAL: NCT05631431
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Curalin As Add-On Therapy in Adults With Type 2 Diabetes Mellitus
Brief Title: Evaluation of Efficacy and Safety of Curalin As Add-On Therapy in Adults With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CuraLife (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Cura-01
Record Dates: First submitted 2021-06-08; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Type2 Diabetes
Keywords: Diabetes; Type 2 Diabetes; placebo; Curalin; CuraLife; Momordica Charantia; Gymnema Sylvestre; Trigonella Foenum Graecum; Curcuma Longa; Emblica Officinalis; Swertia Chirata; Picrorhiza Kurroa; Syzygium Cumini/ Eugenia Jambolana; Cinnamomum Zeylanicum
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Double-blind for 3 months, after 3 months - open-label
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Curalin
- Treatment (Active Comparator)
  Interventions: Dietary Supplement: Curalin

INTERVENTIONS:
Dietary Supplement: Curalin — Curalin capsules, 2 capsules, 3 times a day after meals Placebo: matching placebo capsules, 2 capsules, 3 times a day after meals

SUMMARY:
Evaluation of Efficacy and Safety of Curalin As Add-On Therapy in Adults with Type 2 Diabetes Mellitus

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Curalin As Add-On Therapy in Adults with Type 2 Diabetes Mellitus

ELIGIBILITY:
Diagnosis and Criteria for Inclusion:

Patients may be included in the study if they meet all of the following criteria:

* Written informed consent is obtained.
* Adult patients (18-85 years of age) with Type II diabetes mellitus
* HbA1c at screening is 7.5% - 10%
* Body mass index (BMI)>25
* Stable body weight (±10%) within the 3 months preceding study entry

  • Patients were steadily treated with anti-diabetic medications, such as: GLP-1, Glucophage, DPP-4 inhibitor, or SGLT-2 inhibitor for at least 3 months or more prior to study entry
* The patient must be willing and able to comply with study restrictions and to remain at the clinic for the required duration during the study period, and willing to return to the clinic for the follow-up evaluation as specified in this protocol.

Criteria for Exclusion: Patients will be excluded from participating in this study if they meet 1 or more of the following criteria:

* Patients who have been using Curalin At least once in the past 3 months
* Persons with known sensitivity to any of the components of the Curalin product.
* The patient has any clinically significant uncontrolled medical condition (treated or untreated).
* Patients with renal insufficiency (glomerular filtration rate [GFR]≤30 mL/min/1.73m2)
* Pregnant or lactating women. Women of childbearing potential will be administered a urine pregnancy test at study entry. All study participants will confirm their willingness to use birth control throughout the study.
* Patients deemed by the Investigator as unable to complete study participation.
* Patients currently treated with insulin or those that have been treated with insulin for more than 10 days in the 3 months prior to study entry.

  • Use of medications known to modify glucose metabolism or to decrease the ability to recover from hypoglycemia such as oral, parenteral, local, dermal and inhaled steroids, and immunosuppressive or immunomodulating agents for more than a month prior to study entry, or during the study
* The patient participated in a clinical study (investigational study drug or study device) within 30 days of the study entry
* Life expectancy less than 1 year
* History of stroke, transient ischemic attack, or myocardial infarction within six months prior to screening

  * Patients with uncontrolled hypertension defined as a systolic blood pressure ≥180 mmHg or a diastolic blood pressure ≥100mmHg.
  * Patients who have thyroid-stimulating hormone (TSH) levels >1.5 times the upper limit of normal.
  * Patients with significant liver disease or liver function impairment defined as any of the following; cirrhosis, hepatitis, biliary obstruction with hyperbilirubinemia (total bilirubin >2 times the upper limit of normal) and aspartate aminotransferase (AST) or alanine aminotransferase levels (ALT) >3 times the upper limit of normal.
  * Patients with creatine kinase concentrations > 10 times the upper limit of normal or creatine kinase elevation due to known muscle disease at visit 1 (screening 1)
* Laboratory abnormalities at screening including:
* Potassium > 5.5 mEq/L
* Sodium under 130 mEq/L
* Hemoglobin under 10 g/dl for Women or Under 11 g/dl for man

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
primary objective | 3-6 months
  The primary objective of this study is to evaluate the effect of treatment with Curalin on the change in plasma HbA1c.

CONTACTS AND LOCATIONS:
Locations (4):
- Israel (4):
  - Soroka Medical Center, Beersheba
  - Lin Medical Center, Haifa
  - Herzelia Diebetes Center, Herzliya
  - Ichilov Medical Center, Tel Aviv